CLINICAL TRIAL: NCT01792154
Title: Specular Photomicrograpic Assessment of the Effect of Anti-VEGF Intravitreal Injections on Corneal Thickness and Endothelial Cell Density and Morphology
Brief Title: Measuring Corneal Cells With Specular Microscopy
Status: Completed | Type: Observational
Sponsor: Retina Institute of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: RIH 1011
Record Dates: First submitted 2013-02-11; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Retinal Diseases
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Assess changes in the corneal cell count using Specular Microscopy following tretments with Anti-VEGF injections

DETAILED DESCRIPTION:
Patients with active Wet AMD often receive intraocular Anti-VEGF injections such as Macugen, Lucentis and Avastin on a monthly basis for an extended period of time. While these medications are very effective at controlling the Choroidal Neovascularization associated with this disease, the impact of monthly intravigtreal Anti-VEGF injections on the viability of corneal endothelial cells has yet to be fully characterized. The availability of CESM as a diagnostic test that can be performed quickly and painlessly in the clinic offers a method of tracking corneal endothelial cell count in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Wet Age-related Macular Degeneration
* Receiving monthly intraocular injections of Anti-VEGF medication for at least 3 months
* Age greater than 50 years of age

Exclusion Criteria:

* experiences adverse events

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects of either gender with an age greater than 50 years of age who have been receiving intraocular Anti-VEGF medication every month for at least the past 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Specular Photomicrographic Assessment of the Effect of Anti-VEGF Intravitreal injections on corneal thickness and endothelial cell density and morphology | Baseline, Month 6 and Month 12
  Changes in corneal endothelial cell density and corneal thickness measured by changes in pachymetry and corneal cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Bennett, MD, Principal Investigator — Retina Institute of Hawaii
Locations (1):
- Retina Institute of Hawaii, Honolulu, Hawaii, United States